CLINICAL TRIAL: NCT00682656
Title: Open Label Randomized Study to Assess Safety and Efficacy of Azithromycin Versus Meglumine Antimoniate to Treat Cutaneous Leishmaniasis
Brief Title: Safety and Efficacy of Azithromycin to Treat Cutaneous Leishmaniasis
Acronym: PCL01
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Efficacy issues on test arm
Sponsor: Ana Rabello (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Ana Rabello, Dr. Ana Rabello, Oswaldo Cruz Foundation
Organization: Oswaldo Cruz Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPSH/CPqRR 21/2006
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2011-07

CONDITIONS: Cutaneous Leishmaniasis
Keywords: cutaneous leishmaniasis; azithromycin; N- methyl glucamine
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - N- methyl glucamine (Active Comparator): Glucantime® , max day of 1,215 mg
  Interventions: Drug: Glucantime®
- B - Azithromycin (Experimental): Zithromax ® , one dose 500 mg
  Interventions: Drug: Zithromax ®

INTERVENTIONS:
Drug: Glucantime® — 15mg Sb+5/Kg/day, during 20 days. Maximum dose:15ml/day
  Other Names: meglumine antimoniate
  Arms: A - N- methyl glucamine
Drug: Zithromax ® — Zithromax ®/ Pfizer, 500 mg - 1x day, during 20 days
  Other Names: SELIMAX®
  Arms: B - Azithromycin

SUMMARY:
The adequate treatment of the American tegumentary leishmaniasis is crucial since the disease, differently from the caused by the Old World species, is painful and not self-healing and may lead to the disfiguring mucosal involvement. So far, pentavalent antimony compounds have been considered the treatment of choice for cutaneous leishmaniasis (CL), however, these drugs present high frequency of side effects and important disadvantages as parenteral administration and need for careful renal and cardiac monitoring. Azithromycin is a macrolide antibiotic, non-expensive, largely commercially available that has shown in-vitro and in vivo activity against different species of Leishmania.

The main objective of this study is to evaluate the efficacy and safety of oral azithromycin for the treatment of CL. The efficacy of oral treatment of azithromycin 500 mg/day for 20 days is going to be compared with the standard treatment of intramuscular injections of 20 mg/Kg/day of pentavalent antimonials (Glucantime®) for 20 days in patients with CL from two endemic regions of Brazil: the metropolitan region of Belo Horizonte and Montes Claros (MG)in the southeast Brazil and in Corte de Pedras (Bahia), Northeastern Brazil. The patients follow up lasts for 12 months.

DETAILED DESCRIPTION:
Included a new site (University Estadual de Montes Claros - UNIMONTES) in 7 June 2010. The site was included due the need to achieve more patients. The ANVISA (National Agency of Sanitary Surveillance) approved these site in March 2011 and the start of activities is planned for June 2011.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 14 and younger than 65 years old
* Skin lesions with clinical suggestion of cutaneous leishmaniasis and positive leishmanin skin test(Montenegro test)or parasitological (direct observation of leishmania amastigotes, leishmania in vitro culture from aspirates, histopathological) and molecular(Polymerase Chain Reaction - PCR)samples.
* No use of oral potentially antileishmanial drugs, or topics throughout the term of the current injury.
* Absence of disseminated leishmaniasis.
* Absence of mucosal involvement.
* Agreement to participate in the study and signed the informed consent.

Exclusion Criteria:

* Diabetes mellitus, kidney diseases, liver or cardiac diseases, tuberculosis, malaria.
* Pregnancy
* lactating mothers
* Breast feeding
* Cutaneous lesion with bacterial infection for which antibiotics need to be prescribed
* More than six cutaneous lesions
* Previous history of cutaneous or mucosal leishmaniasis
* Use of drugs with potential pharmacological interactions with antimonials as anti-arrhythmic or tricycle anti-depressives
* Previous intolerance to azithromycin or other macrolides or N-methylglucamine
* Abusive alcohol ingestion according to the CAGE questionnaire

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Proportion of clinically cured patients | at the third month after treatment
  A cure was defined as complete lesion healing and re-epithelialization without inflammatory infiltration and erythema until 90 days after the treatment ended.

SECONDARY OUTCOMES:
Proportion of patients with failure and cured | twelve months after treatment
  Proportion of cured patients at 1, 2, 3, 6, 9 and 12 follow-up after completion of treatment. Mean time to healing.
Occurrence of mucosal lesions after treatment | twelve months after treatment
  Proportion of patients with relapsed or mucosal lesion in 6 months, 9 and 12 follow-up after completion of treatment.
Proportion of patients presenting new lesions | 1st 2nd 3rd 6th 12th month after treatment
  Proportion of patients with new lesions at 1, 2, 3, 6, 9 and 12 follow-up after completion of treatment.
Proportion of adverse events on each treatment group | 1st 2nd 3rd 6th 12th month after treatment.
  Proportion of patients clinical, electrocardiographic and laboratory adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rabello, MD PhD, Principal Investigator — Oswaldo Cruz Foundation; Isabela Ribeiro, MD, Study Director — Drugs for Neglected Diseases
Locations (3):
- Brazil (3):
  - Núcleo de Medicina Tropical University of Brasília - Health Center Corte de Pedras, Presidente Tancredo Neves, Estado de Bahia
  - Centro de Pesquisas René Rachou - Fiocruz, Belo Horizonte, Minas Gerais
  - University Estadual de Montes Claros, Montes Claros, Minas Gerais